CLINICAL TRIAL: NCT02321683
Title: No Mid-term Advantage by Electrochemical Deposition of Hydroxyl-apatite in Cementless Femoral Stems. 5-year RSA and DXA Results From a Randomized Controlled Trial
Brief Title: Evaluation of a New Coating in Cement Less Femoral Stems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Nordsletten (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor-Investigator, Lars Nordsletten, Professor Lars Nordsletten, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO.CR.GH30.
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bonemaster (Experimental): Cement-less femoral stems with electrochemical deposition of hydroxyapatite
  Interventions: Device: Taperloc
- Hydroxyapatite (Active Comparator): Cement-less femoral stems with plasmasprayed hydroxyapatite
  Interventions: Device: Taperloc

INTERVENTIONS:
Device: Taperloc — Femoral stem with electrochemical deposition of hydroxyapatite

SUMMARY:
The purpose of this trial is to evaluate a new method of applying hydroxyapatite coatings on cement-less femoral stems.

DETAILED DESCRIPTION:
60 patients eligible for total hip replacement will be randomized in to two groups, receiving either femoral stems with plasma sprayed hydroxyapatite coating or stems with electrochemically deposited hydroxyapatite. This patients will be followed for at least 5 years. The outcome is evaluated by comparing stability measured by RSA and periprosthetic bone remodeling measured by bone densitometry.

ELIGIBILITY:
Inclusion Criteria:

* non-inflammatory hip arthritis, life expectancy of at least 10 years and hip anatomy allowing the use of standard implants

Exclusion Criteria:

* infection, revision surgery, severe morbidity and obvious bone loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-12; Primary Completion 2005-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Early and intermediate periprosthetic bone remodeling | 5 years
  Bone densitometry measured by DXA
Early and intermediate femoral stem stability | 5 years
  Radiostereometric analysis of femoral stem movements relative to bone

SECONDARY OUTCOMES:
Clinical function | 5 years
  Hip questionares, Harris Hip Score and Oxford Hip Score
Radiographic signs of loosening | 5 years
  Conventional x-ray

REFERENCES:
- [Derived] Flatoy B, Rohrl SM, Boe B, Nordsletten L. No medium-term advantage of electrochemical deposition of hydroxyapatite in cementless femoral stems. 5-year RSA and DXA results from a randomized controlled trial. Acta Orthop. 2016 Feb;87(1):42-7. doi: 10.3109/17453674.2015.1084768. Epub 2015 Sep 12. PMID 26364953